CLINICAL TRIAL: NCT06332313
Title: Comparison of Patient-Controlled Analgesia and Erector Spina Blocks Applied at Different Volumes in Postoperative Pain Management in Retrograde Intrarenal Surgery Operations
Brief Title: Erector Spina Plane Block Volume Comparison
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Boran, associate professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/10/05
Record Dates: First submitted 2024-03-11; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group control (No Intervention): The control group is followed with PCA without a block.
- Group E20 (Active Comparator): Group E20 receive PCA with 20cc volume of ESP block
  Interventions: Procedure: erector spina plane block
- Group E30 (Active Comparator): Group E30 receive PCA with 30 volume of ESP block çevir
  Interventions: Procedure: erector spina plane block

INTERVENTIONS:
Procedure: erector spina plane block — ESP block is a method used to provide postoperative analgesia by injecting local anesthetic between the erector spinae muscle and the transverse process of the vertebra under ultrasound guidance, targeting the dorsal and ventral rami of thoracic and abdominal spinal nerves. The aim of this randomized controlled study is to observe whether there is a difference in tramadol consumption within 24 hours after surgery between patients who undergo RIRS operations at T11 level with different volumes of ESP blocks performed under ultrasound guidance before general anesthesia induction.
  Arms: Group E20; Group E30

SUMMARY:
After obtaining ethical committee approval from Kahramanmaras University Anesthesiology and Reanimation Department and Urology Clinic, 60 patients between 18-65 years old who meet ASA I-II classification criteria with body mass index ≤40 will be informed about this study both verbally and in writing prior to their inclusion in this study using a randomization method according to Helsinki Declaration after obtaining their written consent. Patients who cannot give consent due to any reason or have allergy history against local anesthetics or contraindications for peripheral nerve blocks (local infection,coagulopathy etc.) or psychiatric disorders or receiving antipsychotic drugs will be excluded from this study. Routine preoperative evaluation including age, height, and weight measurements will be performed on all patients at pre-anesthesia clinic.

Patients will be randomized into three groups: Group K, who will receive analgesia with patient-controlled analgesia (PCA) with tramadol only; Group E20, who will receive PCA with 20cc volume of ESP block; and Group E30, who will receive PCA with 30cc volume of ESP block. After standard general anesthesia induction and endotracheal intubation, one of the three analgesic methods will be randomly applied, and the surgery will commence. All patients will receive patient-controlled analgesia. Patients in Group K will not receive any local anesthetic injection. When the patient is transferred to the postoperative care unit, intravenous PCA device will be attached, and pain scores using Visual Analog Scale (VAS), rated from 0 (no pain) to 10 (worst pain ever experienced), at rest and during coughing will be evaluated at 2, 4, 6, 12, 18, and 24 hours postoperatively. The values will be recorded. When the patient experiences pain, analgesic agents will be administered according to the patient-controlled analgesia protocol. The time of first analgesic requirement and total amount of consumed analgesic agent within 24 hours will be recorded. Postoperative QUIPS: Quality Improvement in Postoperative Pain Management questionnaire will be administered, and side effects such as nausea/vomiting or sedation will be noted. Additionally, patient satisfaction regarding these methods and their willingness for repeat surgery or recommendation level on a scale from poor to excellent (very poor/poor/fair/good/excellent)will also be evaluated and recorded

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years old
* ASA I-II classification
* Body mass index ≤40
* Helsinki Declaration after obtaining their written consent
* Patients undergoing Retrograde Intrarenal Surgery

Exclusion Criteria:

* Allergy history against local anesthetics
* Contraindications for peripheral nerve blocks (local infection,coagulopathy etc.)
* Psychiatric disorders or receiving antipsychotic drugs
* Patients with contraindications for spinal anesthesia,
* Coagulopathy,
* Known allergies to the drugs to be used,
* Infection at the site of the procedure,
* Dermatological diseases such as psoriasis that prevent aseptic preparation of the skin at the injection site,
* Septicemia or bacteremia,
* Shock or severe hypovolemia,
* Patients who are not volunteers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-12 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
The aim is to observe the difference in tramadol consumption within the first 24 hours after surgery in 3 groups. | 2, 4, 6, 12, 18, and 24 hours

IPD SHARING:
Plan to Share IPD: No